CLINICAL TRIAL: NCT00396058
Title: Methylphenidats Betydning for motoriskindlæring Hos Patienter Med Apopleksi
Brief Title: The Effect of Methylphenidate on Motor Learning in Stroke Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment of patients proved much too difficult based on the chosen criteria.
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-002554-29
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
The purpose of the study is to determine whether methylphenidate facilitates so called short-term plasticity as measures with transcranial magnetic stimulation, in patients with stroke.

DETAILED DESCRIPTION:
Stroke patients are to be examined with transcranial magnetic stimulation (TMS) before and after a short training session. TMS will be used to demonstrate changes in cortical excitability (motor threshold) and intracortical inhibition and facilitation. The effect of methylphenidate on baseline TMS measures will be evaluated as well as the effect on training induced changes in TMS measures (by comparing baseline and posttraining measures). The patients will be trained on two separate occasions, to compare the effect of Methylphenidate to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Less than two months after first stroke.
* Moderate to light hand paralysis
* Measurable MEP in the abductor pollicis brevis muscle
* Able to read and understand the written information
* Signed informed consent

Exclusion Criteria:

* Epilepsy
* Glaucoma
* Hyperthyroidism
* Cardiac arrythmia
* Known heart disease or angina.
* Metal implants
* Pacemaker
* Pregnancy
* Diastolic BP>100 mmHg
* In treatment with MAO-inhibitor, SSRIs og Ritalin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2006-11; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Training induced changes in Short interval Intracortical Inhibition (SICI).
Training induced changes in Intracortical facilitation (ICF)

SECONDARY OUTCOMES:
Baseline SICI, ICF, and motor threshold compared between methylphenidate and Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jakob U Blicher, MD, Principal Investigator — Hammel neurocenter Aarhus University Hospital Denmark
Locations (2):
- Denmark (2):
  - Department of neurology, Aarhus, Aarhus
  - Hammel neurocenter, Hammel, Hammel